CLINICAL TRIAL: NCT02913430
Title: Treatment of Metastatic Breast Cancer With Fulvestrant Plus Palbociclib or Tamoxifen Plus Palbociclib: A Randomized Pilot Trial With ESR1 Mutation Tested in Circulating Tumor DNA.
Brief Title: Treatment of Metastatic Breast Cancer With Fulvestrant Plus Palbociclib or Tamoxifen Plus Palbociclib
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shannon Puhalla (Other)
Responsible Party: Sponsor-Investigator, Shannon Puhalla, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 16-015
Record Dates: First submitted 2016-09-01; First posted 2016-09-23 (Estimated); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Breast Cancer
Keywords: ESR1 mutation
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Tamoxifen; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): fulvestrant administered 500mg IM Q28 days plus palbociclib125mg/day PO on a 21 days on/7 days off schedule
  Interventions: Drug: Fulvestrant; Drug: Palbociclib
- Arm B (Active Comparator): Tamoxifen is administered orally, at a dose of20mg PO Qdaily plus palbociclib125mg/day PO on a 21 days on/7 days off schedule
  Interventions: Drug: Tamoxifen; Drug: Palbociclib

INTERVENTIONS:
Drug: Fulvestrant — 500mg IM Q28 days
  Arms: Arm A
Drug: Tamoxifen — 20mg PO Qdaily
  Arms: Arm B
Drug: Palbociclib — Tamoxifen or Fulvestrant plus palbociclib125mg/day PO on a 21 days on/7 days off schedule

SUMMARY:
To assess longitudinal changes in allele frequency of ESR1 mutation in plasma in patients treated with Fulvestrant plus palbociclib compared to tamoxifen plus palbociclib

DETAILED DESCRIPTION:
The primary objectives are to assess longitudinal changes in allele frequency of ESR1 mutation in plasma in patients treated with Fulvestrant plus palbociclib compared to tamoxifen plus palbociclib.

Patients with ER+ breast cancer who had 1 to 3 prior lines of endocrine therapy and up to one line of chemotherapy for MBC, excluding fulvestrant and tamoxifen, will be randomized in a 1:1 ratio to receive fulvestrant 500mg IM Q28 days with one extra dose on Day15 of the first cycle (as a loading dose) plus palbociclib 125mg/day PO on a 21 days on/7 days off schedule or tamoxifen 20mg PO daily plus palbociclib 125mg/day PO on a 21 days on/7 days off schedule.

ELIGIBILITY:
For inclusion in the study subjects should fulfill the following criteria:

1. Signed informed consent
2. Patients must have histologically or cytologically confirmed invasive breast cancer that is ER+ (>1% staining) with radiographical or clinical evidence of metastatic disease

   a. Measurable and/or non-measurable disease
3. Prior therapies:

   1. Patients must have previously received an aromatase inhibitor in the adjuvant, neo-adjuvant or metastatic setting.
   2. Patients must have previously received palbociclib in the adjuvant, neo- adjuvant or metastatic setting. If patient is currently taking palbociclib at time of screening for the trial they may continue taking palbociclib.
   3. The minimum duration of AI in the adjuvant setting is 2 years.
   4. There is no minimum duration of AI in the metastatic setting or neoadjuvant setting.
   5. Patients may have been previously treated with an mTOR inhibitor or other investigational agent in addition to an aromatase inhibitor.
   6. Prior treatment with tamoxifen is allowed in the adjuvant setting provided that it was followed by a minimum of 2 years of an AI.
4. Brain metastasis is allowed if previously treated, stable and off steroids for a minimum of 56 days
5. Age > 18 years
6. Male or female breast cancer is allowed
7. Patients may be pre- or post-menopausal; pre-menopausal patients must be on ovarian suppression and must be adequately suppressed on LHRH agonists with estradiol levels in the post-menopausal range

   a. Premenopausal patients cannot be pregnant and must agree to adequate birth control in addition to ovarian suppression. Agreement by the patient and/or partner to use highly effective, nonhormonal form of contraception or two effective forms of non-hormonal contraception. Contraception use should continue during the duration of study treatment and for at least 6 months after the last dose of study treatment.
8. ECOG performance status 0-2
9. Adequate bone marrow function as indicated by the following, within 14 days of enrollment:

   1. ANC ≥ 1500 cells/mm3
   2. Platelets ≥ 100,000 cells/ mm3
   3. Hemoglobin ≥ 9 g/dL
10. Adequate liver function, as indicated by the following, within 14 days of enrollment.

    1. Total bilirubin 1.5 upper limit of normal (ULN)
    2. AST 1.5 ULN
    3. ALT ≤ 2.5 ULN
    4. Alkaline phosphatase ≤ 2.5 ULN with the following exception; ALP ≤ 5× ULN in patients with bone metastases.
11. Adequate hemostatic function as determined by PT, INR and aPTT < 1.5× ULN (unless on therapeutic coagulation, in which case the adequate level of anticoagulation will be determined by the investigator).
12. Adequate renal function, as indicated by creatinine ≤ 1.5 ULN.

Subjects should not enter the study if any of the following exclusion criteria are fulfilled

1. Prior therapy exclusions:

   1. Prior therapy with fulvestrant
   2. Prior therapy with tamoxifen in the metastatic setting
   3. More than 3 prior lines of endocrine therapy in the metastatic setting
   4. More than one prior line of chemotherapy in the metastatic setting
2. Washout of 2 weeks is required for aromatase inhibitors; washout of 4 weeks is required for, everolimus or other biological agents with the exception of Palbociclib.
3. Patients must not be receiving any other investigational agent.
4. Patients with symptomatic, untreated CNS metastases are not eligible.
5. Patients may not have significant concurrent illness, infection, pregnancy or lactation
6. Patients must not have a different active malignancy, except for skin basal cell carcinoma, skin squamous cell carcinoma and cervical intraepithelial neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Puhalla, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients
Groups:
- Fulvestrant + Palbociclib: Fulvestrant: 500mg IM Q28 days
  Palbociclib: 125mg/day PO on a 21 days on/7 days off schedule
- Tamoxifen + Palbociclib: Tamoxifen: 20mg PO Q-daily
  Palbociclib: 125mg/day PO on a 21 days on/7 days off schedule
Period: Overall Study
Arm/Group | Fulvestrant + Palbociclib | Tamoxifen + Palbociclib
Started | 5 | 2
Completed | 5 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant + Palbociclib | Tamoxifen + Palbociclib | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.00 (14.32) | 69.50 (4.95) | 66.29 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Status (at study entry) [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance measures a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. Scoring ranges from 0 to 5 and are as follows: 0 = Normal Activity, asymptomatic, 1 = Symptomatic, fully ambulatory, 2 = Symptomatic; in bed < 50% of time, 3 = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours, 4 = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair, and, 5 = Death
  Participants
    ECOG = 0 | 3 | 1 | 4
    ECOG = 1 | 1 | 1 | 2
    ECOG = 2 | 1 | 0 | 1
    ECOG = 3 | 0 | 0 | 0
    ECOG = 4 | 0 | 0 | 0
    ECOG = 5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The duration of time from time of randomization to time of progression or death, whichever occurs first. Disease progression (PD) as defined by RECIST v1.1: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The progression of non-target lesions or the appearance of one or more new lesions is also considered progression.
  PFS for a subject without an event will be censored on the date of last tumor assessment. If an interval of 6 months passes without a tumor assessment, PFS will be censored at the time of the earlier tumor assessment, even if an event (progressive disease or death) is later observed.
Time Frame: Up to 3 years and 351 days
Population: Treated patients that were radiologically evaluable.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant + Palbociclib | Tamoxifen + Palbociclib
Number analyzed (Participants) | 5 | 2
months | 4.131147 [1.672131 to NA] — Upper bound of confidence interval not reached. Insufficient number of participants with events. | NA [NA to NA] — Confidence interval NOT determined. Insufficient number of participants with events.

2. Secondary Outcome: Best Overall Response (BOR)
Description: The number of patients experiencing Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD) per RECIST v1.1; Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1): (CR) is disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; (SD) is neither sufficient decrease (target lesions) to qualify as a PR or sufficient increase to qualify as PD. Incomplete Response/Stable Disease (SD) is the persistence of one or more non-target lesions. (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions compared to baseline sum of target lesions, or any new lesions. It also includes the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 5 years
Population: Treated patients that were radiologically evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant + Palbociclib | Tamoxifen + Palbociclib
Number analyzed (Participants) | 5 | 2
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Stable Disease (SD) | 3 | 2
  Progressive Disease (PD) | 2 | 0

3. Secondary Outcome: 6-Month Clinical Benefit Rate (CBR)
Description: The number of patients experiencing Complete Response (CR), Partial Response (PR), or Stable Disease (SD) per RECIST v1.1; Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1): (CR) is disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; (SD) is neither sufficient decrease (target lesions) to qualify as a PR or sufficient increase to qualify as PD. Incomplete Response/Stable Disease (SD) is the persistence of one or more non-target lesions.
Time Frame: Up to 6 months
Population: Treated patients that were radiologically evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant + Palbociclib | Tamoxifen + Palbociclib
Number analyzed (Participants) | 5 | 2
Participants | 2 | 1

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: as for outcome 3
Time Frame: Up to 5 years
Population: Treated patients that were radiologically evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant + Palbociclib | Tamoxifen + Palbociclib
Number analyzed (Participants) | 5 | 2
Participants | 3 | 2

5. Secondary Outcome: Overall Survival (OS)
Description: The median length of time from the start of treatment that patients remain alive.
Time Frame: Up to 5 years
Population: All enrolled patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant + Palbociclib | Tamoxifen + Palbociclib
Number analyzed (Participants) | 5 | 2
months | NA [11.77049 to NA] — Insufficient number of participants with event. | 18.75410 [18.75410 to NA] — Insufficient number of participants with event.

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Arm/Group | Fulvestrant + Palbociclib | Tamoxifen + Palbociclib
All-Cause Mortality (participants affected / at risk) | 1/5 | 1/2
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/2
Other Adverse Events (participants affected / at risk) | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Palbociclib (N=5) | Tamoxifen + Palbociclib (N=2)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 | 0
White blood cell decreased (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Palbociclib (N=5) | Tamoxifen + Palbociclib (N=2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 1
General disorders and administration site conditions (General disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Pain (General disorders) | 2 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 1 | 0
Flu like symptoms (General disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nervous system disorders - Other (Nervous system disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Psychiatric disorders - Other (Psychiatric disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 1
White blood cell decreased (Investigations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT02913430/Prot_SAP_000.pdf